CLINICAL TRIAL: NCT00343044
Title: Phase II Study of Weekly Topotecan With Bevacizumab in Platinum Resistant Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancers
Brief Title: Ph II Study of Wkly Topotecan + Bevacizumab in Plat. Resistant/Recurrent Gyn Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Beth Edelheit, Thomas Malpass, MD, Kathryn McGonigle, MD, Benaroya Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3040200; AVF3648s (Other: GSK)
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: platinum resistant ovarian cancer; recurrent ovarian cancer; platinum resistant cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Topotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects received standard topotecan with the addition of bevacizumab. Cycles were 28 days and continued until toxicity, progression or subject wish to discontinue treatment. Topotecan administered 4 mg/m2 IV on days 1, 8 and 15 and bevacizumab IV 10 mg/kg, days 1 and 15 of each cycle.
  Interventions: Drug: Topotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Topotecan — Topotecan administered days 1, 8, and 15 of each 28 day cycle. Dose was 4 mg/m2 administered IV.
  Other Names: Hycamtin
Drug: Bevacizumab — bevacizumab administered IV 10 mg/kg, days 1 and 15 of 28 day cycle.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the clinical safety and toxicity of intravenous bevacizumab (Days 1 and 15 of a 28 day cycle) in combination with weekly topotecan (Days 1, 8, 15 of a 28 day cycle) in patients with platinum resistant recurrent ovarian, fallopian tube and primary peritoneal cancer.

DETAILED DESCRIPTION:
This study is designed as a Phase 2 study. There are no published data on the toxicity of the combination of bevacizumab and topotecan therapy. Based on data combining bevacizumab with other chemotherapy agents in non-gynecologic solid tumors, it is not likely that the toxicity of the combination of the two drugs will be greater than the individual toxicities of each drug. The toxicities of each of these agents is quite different. Specifically the toxicity of this combination will be studied using the dose of bevacizumab used in previous phase II studies of ovarian cancer, e.g. an equivalent of 5 mg/kg weekly with treatments given at least every 3 weeks. In our study, since topotecan will be given weeks 1,2 and 3 of an every 4 week cycle, it is convenient to give bevacizumab 10 mg/kg IV every other week.

ELIGIBILITY:
Inclusion Criteria:

* must have received primary taxane and platinum-based chemotherapy and no more than 1 other chemotherapy regimen
* must have platinum resistant disease(defined as recurrence within 6 months of receiving platinum based chemotherapy, first or second line)
* must have measurable disease (greater than 20mm by conventional techniques or 10mm by spiral CT) OR elevated CA-125 (> 100 on two occasions at least one week apart
* performance status greater than or equal to 70%

Exclusion Criteria:

* prior treatment with anti-angiogenesis agent
* treatment with > 2 cytotoxic regimens (including primary platinum and taxane chemotherapy)
* evidence of other malignancy within 3 years of study enrollment
* history of abdominal fistula, grade 4 bowel obstruction or gastrointestinal perforation
* history of intra-abdominal abscess with 6 months prior to day 0
* pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn McGonigle, MD, Principal Investigator — Virginia Mason Medical Center
Locations (2):
- United States (2):
  - Virginia Mason Medical Center, Seattle, Washington
  - Puget Sound Oncology Consortium (PSOC), Seattle, Washington

REFERENCES:
- [Result] McGonigle KF, Muntz HG, Vuky J, Paley PJ, Veljovich DS, Greer BE, Goff BA, Gray HJ, Malpass TW. Combined weekly topotecan and biweekly bevacizumab in women with platinum-resistant ovarian, peritoneal, or fallopian tube cancer: results of a phase 2 study. Cancer. 2011 Aug 15;117(16):3731-40. doi: 10.1002/cncr.25967. Epub 2011 Feb 24. PMID 21815133
- See also: Benaroya Research Institute's homepage with listings of clinical trials — http://www.benaroyaresearch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled from August 2006 to November 2008, in the medical oncoogy practices at Virginia Mason Medical Center and the Puget Sound Oncology Consortium in Seattle, WA.
Pre-assignment Details: Women had advanced or recurrent epithelial ovarian, peritoneal, or fallopian tube cancer. Enrollment was restricted to women who had received a maximum of two prior chemotherapy regimens, with at least one prior primary taxane and platinum-based therapy.
Groups:
- Combined Weekly Topotecan and Biweekly Bevacizumab: Treatment was administered in 28 day cycles, with IV bevacizumab 10 mg/kg given on days 1 and 15 and IV topotecan 4 mg/m2 given on days 1 and 8. Treatment was continued until progressive disease defined by RECIST, symptomatic deterioration related to clinical progression, excessive toxicity. Dose reductions of bevacizumab were not permitted.
Period: Overall Study
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival(PFS)was measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with measurable disease. For patients with nonmeasurable disease, cancer antigen (CA-125) levels were used to determine response according to Rustin criteria. Progression-free survival was defined as number of months after beginning study treatment until progressive disease or death, respectively.
Time Frame: PFS and OS were defined as the number of months after commencing study treatment until progressive disease or death.
Population: This was determined assuming a median progression free survival of 9 months and an analysis calculating the sample size at which the narrowing of its 95% confidence interval became greater than .20 for every 2 patients added. Progression free survival and overall survival were estimated by using the Kaplan Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Number analyzed (Participants) | 40
months
  All participants | 7.8 [3 to 9.4]
  One prior regimen (n=21) | 2.8 [2.3 to 7.2]
  Two prior regimens (n=19) | 10.9 [7.1 to 14.7]
Statistical Analysis 1: Comparison: Combined Weekly Topotecan and Biweekly Bevacizumab; Planned enrollment of 40 patients was determined assuming a median progression free survival (PFS) of 9 months (based on a median PFS of 7.2 months for low-dose, metronomic cyclophosphamide plus bevacizumab in a phase 2 study) and an analysis calculating the sample size at which the narrowing of its 95% confidence interval (CI) became greater than .2 for every 2 patients added. Progression free survival was estimated using the Kaplan-Meier method; Test type: Superiority or Other; p = .08, Log Rank — Standard statistical methods (log-rank tests) were used in post hoc analyses that compared efficacy parameters in patients who received 1 vs 2 prior treatment regimens

2. Secondary Outcome: Evaluation of Overall Survival
Description: Overall survival was defined as the number of months after commencing study treatment to death.
Time Frame: PFS and OS were defined as the number of months after commencing study treatment until progressive disease or death.
Population: The planned enrollment of 40 participants was determined using a median PFS of 9 months (based on a median PFS of 7.2 months in a previous trial).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Number analyzed (Participants) | 40
months
  All Participants | 16.6 [12.8 to 22.9]
  One Prior Regimen (n=21) | 12.8 [9.0 to 14.9]
  Two Prior Regimens (n=19) | 22.9 [16.6 to 22.9]
Statistical Analysis 1: Comparison: Combined Weekly Topotecan and Biweekly Bevacizumab; Overall survival(OS)was estimated using the Kaplan-Meier method; Test type: Superiority or Other; p = .02, Log Rank — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate
Description: RECIST criteria
Time Frame: Response
Measure: Number; unit: participants
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Number analyzed (Participants) | 40
participants | 10

4. Secondary Outcome: Number or Participants With Toxicity
Time Frame: measured at each treatment cycle
Measure: Number; unit: participants
Arm/Group | Combined Weekly Topotecan and Biweekly Bevacizumab
Number analyzed (Participants) | 40
participants | 40

ADVERSE EVENTS:
Time Frame: Adverse event collecting occurred from first subject enrolled through January 31, 2010.
Description: All patients had been previously treated with platinum (carboplatin or cisplatin) and a taxane (paclitaxel or docetaxel. Toxicity was generally mild or moderate. No treatment related death occurred.
Groups:
- Arm 1: Patients (N=40)
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=40)
Pain (General disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=40)
Neutropenia (Blood and lymphatic system disorders) | 22 (22)
Anemia (Blood and lymphatic system disorders) | 19 (19)
Leukopenia (Blood and lymphatic system disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13)
Fatigue (General disorders) | 20 (20)
Pain (General disorders) | 18 (18)
Nausea/Vomiting/Diarrhea (Gastrointestinal disorders) | 18 (18)
infection (Infections and infestations) | 16 (16)
Depression (Psychiatric disorders) | 3 (3)
Hypertension (Cardiac disorders) | 12 (12)
GGT increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Venous thrombosis (Vascular disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alkaline phosphatase (Investigations) | 2 (2)
Aspartate aminotransferase (Investigations) | 1 (1)
Alanine aminotransferase (Investigations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No